CLINICAL TRIAL: NCT01047280
Title: Use of Conjugated Linoleic Acid as a Nutraceutical for Weight Loss in Humans
Acronym: CLA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Peter J Jones, PhD, Richardson Centre for Functional Foods and Nutraceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B2005:183
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-12

CONDITIONS: Body Weight; Body Composition; Hyperlipidemia; Inflammation; Oxidative Stress
Keywords: Conjugated linoleic acid; Body weight; Body composition; Blood lipid profile; Body inflammatory and oxidative status
MeSH Terms: conditions — Body Weight; Hyperlipidemias; Inflammation | interventions — Safflower Oil; CD2 Antigens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Safflower oil (Placebo Comparator): This arm of the study constitutes the control phase
  Interventions: Dietary Supplement: Safflower oil
- Clarinol G-80® (Experimental)
  Interventions: Dietary Supplement: Clarinol G-80 ® treatment
- G-c9, t11 (Experimental)
  Interventions: Dietary Supplement: G-c9, t11

INTERVENTIONS:
Dietary Supplement: Clarinol G-80 ® treatment — dietary supplement of 3.5g/day 50-50 mixture of t10, c12 and c9, t11 CLA. In addition, the amount of mixed natural tocopherols is 5mg/g (0.05%).
  Arms: Clarinol G-80®
Dietary Supplement: Safflower oil — 3.5 g/d of safflower oil
  Arms: Safflower oil
Dietary Supplement: G-c9, t11 — 3.5 g/day of c9, t11 CLA
  Arms: G-c9, t11

SUMMARY:
The purpose of the study is to examine how a naturally occurring fat found in meats, such as beef and lamb and milk, called conjugated linoleic acid (CLA), will affect your body weight and body fat content, blood fat levels, as well as selected safety parameters. The CLA will be supplemented in an oil form and will be added to solid foods as provided by the metabolic kitchen at the Richardson Centre for Functional Foods and Nutraceuticals (RCFFN).

DETAILED DESCRIPTION:
In order to investigate the effectiveness of CLA on body weight and composition, as well as blood lipids, a double-blinded, 3-phase crossover trial will be conducted in moderately overweight (BMI=25-40 kg/m2), borderline hypercholesterolemic (LDL-C ≥ 2.5 mmol/L) men between the ages of 18-60 years. During three 8-week phases separated by 4-week washout periods, and under supervision to ensure compliance, 28 subjects will consume in random order (i) Control: 3.5 g/d of safflower oil, (ii) Clarinol G-80®: 3.5 g/d of 50:50 mixture of t10, c12 and c9, t11 CLA and (iii) c9, t11: 3.5 g/day of c9, t11 CLA. Body weight, fat mass and lean body mass will be measured at beginning and end of each phase by dual energy X-ray absorptiometry (DEXA). Baseline and endpoint blood samples will collected to determine blood lipid profile, and different safety parameters, including insulin sensitivity (HOMA-IR index), and concentrations of inflammatory (hs-CRP, TNF-α, IL-6) and oxidative (Oxidized-LDL) biomarkers. Effect of CLA consumption on fatty acid oxidation will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Study subjects will be defined as overweight or obese, hyperlipidemic males, with a LDL-C level of greater than 2.5 mmol/L.Subjects will be between 18-60 years old and must have a body mass index (BMI) of 25-36 kg/m2. Subjects with thyroid diseases will be included in the study as long as they have been shown to be stable in response to their medications and thyroid therapy will have to be maintained at a stable dose throughout the study.

Exclusion Criteria:

1. subjects taking medications and/or natural health products known to affect lipid metabolism (cholestyramine, colestipol, niacin, clofibrate, gemfibrozil, probucol, HMG CoA reductase inhibitors, high dose dietary supplements or fish oil capsules (> 4 g/day), guggul, lecithin, evening primrose oil within the last six months. In addition subjects will no be allowed to consume any of these medications during the study;
2. subjects who have taken plant sterol supplements within the past six weeks and consume plant sterol supplements during the trial;
3. subjects who currently have diabetes, kidney, heart or liver disease or have had any of these diseases at any time during the past 3 months. In addition any development of diabetes mellitus, kidney, heart or liver disease during the trial will lead to exclusion from the trial;
4. subjects who smoke or consume large amounts of alcohol (> 2 drinks/day);
5. subjects who have any major food allergies or are vegetarian;
6. subjects that use natural or pharmaceutical weight loss supplements or products known to affect lipid metabolism at the beginning and end of each treatment period as well as the washout periods;
7. subjects who are sensitive to the Asteraceae/Compositae family (e, g., ragweed, marigolds, daisies).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Changes in body weight, body fat mass, and lean body mass | At baseline and endpoint of each phase

SECONDARY OUTCOMES:
Changes in inflammation and oxidation markers | At baseline and endpoint of each phase

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, Ph.D., Principal Investigator — University of Manitoba

REFERENCES:
- [Derived] Joseph SV, Jacques H, Plourde M, Mitchell PL, McLeod RS, Jones PJ. Conjugated linoleic acid supplementation for 8 weeks does not affect body composition, lipid profile, or safety biomarkers in overweight, hyperlipidemic men. J Nutr. 2011 Jul;141(7):1286-91. doi: 10.3945/jn.110.135087. Epub 2011 May 18. PMID 21593349